CLINICAL TRIAL: NCT00621647
Title: A Multicenter, Double-Blind, Randomized, Comparison of the Efficacy and Safety of Quetiapine Fumarate (SEROQUEL) and Placebo in the Treatment of Agitation Associated With Dementia.
Brief Title: Seroquel- Agitation Associated With Dementia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans Eriksson / Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 5077US/0046; D1446L00002
Record Dates: First submitted 2008-02-06; First posted 2008-02-22 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Alzheimer's Disease; Vascular Dementia
Keywords: Seroquel; dementia; agitation symptoms; Alzheimer's disease; vascular dementia; quetiapine fumarate
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Dementia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 1st fixed dose
  Interventions: Drug: Quetiapine Fumarate
- 2 (Experimental): 2nd fixed dose
  Interventions: Drug: Quetiapine Fumarate
- 3 (Sham Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine Fumarate
  Other Names: Seroquel
  Arms: 1
Drug: Quetiapine Fumarate
  Arms: 2
Drug: Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to determine how safe and effective Seroquel (quetiapine fumarate) is compared to placebo (a non-drug tablet) for a period of up to 10 weeks in the treatment of agitation symptoms in nursing home or assisted care residents.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of dementia compatible with probable or possible Alzheimer's disease (AD)
* Subjects exhibit inappropriate verbal, vocal, or motor activity that requires treatment with an antipsychotic medication in addition to or beyond behavioural modification therapy
* Subject must have a score of at least 14 on the PANSS

Exclusion Criteria:

* Current or past symptoms for schizophrenia, schizoaffective disorder, or bipolar disorder
* Symptoms of agitation that are caused by another general medical condition or direct physiological effects of a substance
* Failure to respond on 2 occasions to an adequate regimen of atypical antipsychotic medications for the treatment of agitation and/or aggression

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2002-09; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of 2 fixed doses of quetiapine compared with placebo | Twice weekly

SECONDARY OUTCOMES:
To assess the efficacy of quetiapine compared with placebo | Twice weekly